CLINICAL TRIAL: NCT06235216
Title: A Multicenter, Open Label, Two Cohort, Single Arm, Phase II Study to Evaluate the Efficacy and Safety of the Anti-TROP2 Antibody-drug Conjugate Sacituzumab Govitecan in Patients With Advanced Differentiated and Anaplastic Thyroid Neoplasms.
Brief Title: Sacituzumab govitEcan in THYroid Cancers
Acronym: SETHY
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Grupo Espanol de Tumores Neuroendocrinos (Other)
Collaborators: MFAR (Other); Gilead Sciences (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GETNE T2318; 2023-504898-20 (EudraCT Number)
Record Dates: First submitted 2024-01-23; First posted 2024-01-31 (Actual); Last update posted 2024-11-01 (Actual); Status verified 2024-10

CONDITIONS: Differentiated Thyroid Cancer; Anaplastic Thyroid Cancer
Keywords: TROP-2; sacituzumab govitecan; Antibody-drug conjugate; SN-38
MeSH Terms: conditions — Thyroid Carcinoma, Anaplastic | interventions — sacituzumab govitecan

STUDY DESIGN:
Intervention Model Description: two cohorts of patients
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Experimental (Experimental): Sacituzumab govitecan (10 mg/kg) administered intravenously on Days 1 and 8 of a 21-day cycle. Patients will be treated until progression, death, study withdrawal, or unacceptable toxicity.
  Interventions: Drug: Sacituzumab govitecan

INTERVENTIONS:
Drug: Sacituzumab govitecan — Dose of 10 mg/kg intravenously
  Other Names: Trodelvy

SUMMARY:
SETHY is a prospective, multicohort, phase II, single-arm, non-randomized, non-blinded, investigator-initiated study of sacituzumab govitecan in patients with advanced or metastatic radioactive-iodine refractory differentiated thyroid carcinoma (DTC) or anaplastic thyroid carcinoma (ATC).

The main hypothesis is that treatment with sacituzumab govitecan, a anti-Trophoblast cell surface antigen 2 (TROP-2), could be an effective treatment option for patients with either differentiated and anaplastic thyroid neoplasms because TROP-2 is highly expressed at the membrane of DTC and ATC.

DETAILED DESCRIPTION:
The trial will enroll competitively up to 21 patients per cohort. The study will enroll the first 12 patients within the cohort and monitor for response. If no confirmed response is documented the cohort will be closed. If there is one or more confirmed responses reported that cohort will be expanded up to the expected 21 patients. All patients, male or female, ≥ 18 years, with ECOG PS 0-1. Cohort 1 will include patients with advanced radioactive-iodine refractory DTC who progressed to previous TKIs (including but not limited to lenvatinib, sunitinib or cabozantinib) and cohort 2 will include patients with advanced or metastatic ATC who may be on first-line or progressed to a previous systemic treatment. Patients will have not received previously chemotherapy, biologics, investigational agents, and/or antitumor treatment with immunotherapy that are not completed 2 weeks before first dose of study treatment (See Section 6 for further detail on eligibility).

All enrolled patients will receive sacituzumab govitecan (10 mg/kg intravenously) on Days 1 and 8 of a 21-day cycle. Patients will be treated until progression, death, study withdrawal, or unacceptable toxicity. Sacituzumab govitecan is administered intravenously as a slow infusion as described below.

Dosing is based on the patient's body weight on Day 1 of each cycle (or at each dosing day if change in body weight is >10% or if required by institutional policy). Sacituzumab govitecan at 10 mg/kg will be the highest assigned dose. Dose reductions and delays will be allowed.

All patients will undergo periodic tumor assessments by CT or MRI scan every 12 weeks ± 14 days (3 months), and blood monitoring of tumor markers (i.e. thyroglobulin if applicable) every 12 weeks ± 3 days (3 months) from the start of study treatment until progression or patient withdrawal.

ELIGIBILITY:
Inclusion Criteria:

1. Institutional Review Board (IRB)/Independent Ethics Committee (IEC) approved written informed consent.
2. Patient is ≥ 18 years of age.
3. Patient has histologically confirmed metastatic or locally advanced unresectable radioactive-iodine refractory differentiated thyroid cancer (cohort A) or anaplastic thyroid carcinoma (cohort B).
4. Prior therapy in each cohort:

   1. Cohort A: Patients must have experienced progression on at least one previous treatment line with approved systemic therapies (Sorafenib, Lenvatinib or Cabozantinib) and a maximum of 3 prior systemic therapies.
   2. Cohort B: Patients should be included in first-line setting or after failure of any systemic therapy (up to 1 prior treatment lines).
5. Patient has radiographically documented and measurable metastatic or locally advanced disease at baseline.
6. An archival tumor tissue sample should be available for submission to the central laboratory for translational studies. If an archival tumor tissue sample is not available, a new biopsy tissue sample should be provided. No central pathological review will be needed to include the patient in the trial.
7. Patient has Eastern Cooperative Oncology Group (ECOG) performance status of 0 or 1.
8. The following baseline laboratory data without transfusional support:

   1. Neutrophil count (ANC) ≥ 1,500/mm3.
   2. Platelet count ≥ 100 × 109/L.
   3. Hemoglobin ≥ 9 g/dL.
   4. Serum bilirubin ≤ 1.5 × upper limit of normal (ULN). Note: patients with Gilbert's disease are excluded.
   5. Serum albumin > 3 g/dL.
   6. Creatinine clearance (CrCl) ≥ 60 mL/min as estimated by the Cockroft-Gault formula or as measured by 24 hour urine collection (GFR can also be used instead of CrCl).
   7. Alanine aminotransferase (ALT) and aspartate aminotransferase (AST) ≤ 2.5 × ULN or ≤ 5 xULN for patients with liver metastases.
9. Female patients must either:

   1. Be of nonchildbearing potential:

      I)Postmenopausal *(defined as at least 1 year without any menses) prior to screening , or II) Documented surgically sterile (e.g.hysterectomy, bilateral salpingectomy, bilateral oophorectomy, or bilateral tubal occlusion).

      *Those who are amenorrheic due to an alternative medical cause are not considered postmenopausal and must follow the criteria for childbearing potential subjects.

      OR
   2. If of childbearing potential:

   I) Agree not to try to become pregnant during the study and for at least 6 months after the final study drug administration, II) And have a negative urine or serum pregnancy test within 7 days prior to Day 1 (females with false positive results and documented verification of negative pregnancy status are eligible for participation), III) And if heterosexually active, agree to abstinence (if in line with the usual preferred lifestyle of the patient) or consistently use a condom plus 1 form of highly effective birth control per locally accepted standards starting at screening and throughout the study period and for at least 6 months after the final study drug administration.
10. Female patients must agree not to breastfeed or donate ovules starting at screening and throughout the study period, and for at least 6 months after the final study drug administration.
11. Male patients must not donate sperm starting at screening and throughout the study period, and for at least 6 months after the final study drug administration.
12. Male patients with a partner with childbearing potential, or who is pregnant or breastfeeding must agree to abstinence or use a condom plus 1 form of highly effective birth control throughout the study period and for at least 6 months after the final study drug administration.
13. Patient agrees not to participate in another interventional study while on treatment in the present study.

Exclusion Criteria:

1. Patient has central nervous system (CNS) metastases.
2. Patient has ongoing clinically significant toxicity (Grade 2 or higher with the exception of alopecia) associated with prior treatment (including systemic therapy, radiotherapy or surgery).

   Note: if patients received major surgery, they must have recovered adequately from the toxicity and/or complications from the intervention prior to starting therapy.
3. Patient has a history of another malignancy within 3 years before the first dose of study drug, or any evidence of residual disease from a previously diagnosed malignancy.

   Note: Patients with non melanoma skin cancer, curatively treated localized prostate cancer, or carcinoma in situ of any type (if complete resection was performed) are allowed.
4. Patient has known active Hepatitis B or active hepatitis C:

   1. Patients who test positive for hepatitis B surface antigen (HBsAg). Patients who test positive for hepatitis B core antibody (anti-HBc) will require HBV DNA by quantitative polymerase chain reaction (PCR) for confirmation of active disease.
   2. Patients who test positive for HCV antibody. Patients who test positive for HCV antibody will require HCV RNA by quantitative PCR for confirmation of active disease. Patients with a known history of HCV or a positive HCV antibody test will not require a HCV antibody at screening and will only require HCV RNA by quantitative PCR for confirmation of active disease.
   3. Patients who test positive for HIV antibody.
5. Patient has a known history of human immunodeficiency virus (HIV) infection (HIV 1 or 2) with detectable viral load OR taking medications that may interfere with SN-38 metabolism.
6. Patient has documented history of a cerebral vascular event (stroke or transient ischemic attack), or the following criteria for cardiac disease:

   1. Myocardial infarction or unstable angina pectoris within 6 months of enrollment.
   2. History of serious ventricular arrhythmia (ie, ventricular tachycardia or ventricular fibrillation), high-grade atrioventricular block, or other cardiac arrhythmias requiring antiarrhythmic medications (except for atrial fibrillation that is well controlled with antiarrhythmic medication); history of QT interval prolongation.
   3. New York Heart Association (NYHA) class III or greater congestive heart failure or left ventricular ejection fraction of < 40%.
7. Known history of clinically significant active COPD, or other moderate-to-severe chronic respiratory illness present within 6 months prior to the first dose of study drug.
8. Patients with active chronic inflammatory bowel disease (ulcerative colitis, Crohn disease) and patients with a history of gastrointestinal obstruction or perforation within 6 months of enrollment.
9. Patient has uncontrolled hypertension or diabetes.
10. Patient has radiotherapy or major surgery within 4 weeks prior to the first dose of study drug.
11. Patients has received a live vaccine within 30 days, or antibiotics within one week prior to the first dose of study drug.
12. Patient has had chemotherapy, biologics, investigational agents, and/or antitumor treatment with immunotherapy that is not completed 2 weeks prior to the first dose of study drug.

    Note: Patients participating in observational studies are eligible.
13. Patient has previously received topoisomerase 1 inhibitors.
14. Patient has known hypersensitivity to sacituzumab govitecan or to any excipient contained in the drug formulation.
15. Patient has other underlying medical conditions that, in the opinion of the investigator, would impair the ability of the patient to receive or tolerate the planned treatment and follow-up.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Estimated)
Dates: Start 2024-09-13 (Actual); Primary Completion 2027-12 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
Objective response rate (ORR) | Throughout the study period, approximately 42 months since the inclusion of first patient
  percentage/proportion of patients with confirmed complete response (CR) or partial response (PR) as their overall best response throughout the study period. Objective responses will be assessed locally by the investigator according to RECIST, version 1.1

SECONDARY OUTCOMES:
Disease control rate (DCR) | Throughout the study period, approximately 42 months since the inclusion of first patient
  Percentage/proportion of patients with complete response (CR) or partial response (PR), according to ORR definition for the trial, or maintained stable disease (SD) as their overall best response, assessed by imaging follow-up (CT scan/MRI) and RECIST 1.1 criteria. Stable disease should be maintained for at least 4 months to be considered as a CBR event.
Duration of response (DoR) | Throughout the study period, approximately 42 months since the inclusion of first patient
  Time from first confirmed response (CR or PR), according to ORR definition for the trial, to the date of the documented PD as determined using RECIST 1.1 criteria or death due to any cause, whichever occurs first. Those patients with response and without PD or death event will be censored on the date of their last tumor assessment.
Progression-free survival (PFS) | Throughout the study period, approximately 42 months since the inclusion of first patient
  Time from first dosing date to the date of confirmed PD according to RECIST 1.1. Patients alive and free of events at the date of the analysis will be censored at their last known tumor assessment. Patients who start a new treatment line without progression will be censored on the date of first dose of the subsequent anticancer treatment.
Overall survival (OS) | Throughout the study period, approximately 42 months since the inclusion of first patient
  Time elapsed from the first dose of study treatment until death from any cause. We will assess the median OS, estimated by Kaplan-Meier. Patients alive and free of events at the date of the analysis will be censored at their last known contact. Survival will be assessed by recording patient status at each visit. Long term follow up to be performed at least every 6 months.
Safety profile | Throughout the study period, approximately 42 months since the inclusion of first patient
  Percentage/proportion of patients that experience adverse events classified by their type, severity and seriousness according to the National Cancer Institute's Common Toxicity criteria (NCI-CTCAE v5.0) scoring system.
Patient self-reported quality of life (QoL) | Throughout the study period, approximately 42 months since the inclusion of first patient
  Assessed at baseline and every 12 weeks until progression through the EORTC QLQ-C30 questionnaire. The questionnaire is a validated tool composed of 30 questions or items that assess QoL in relation to physical, emotional, social aspects. The questionnaire is structured in 5 functional scales (physical functioning, daily activities, emotional functioning, cognitive functioning and social functioning), 3 symptom scales (fatigue, pain and nausea, vomiting), 1 global health status scale, and 6 independent items (dyspnea, insomnia, anorexia, constipation, diarrhea and economic impact). Values between 1 and 4 (1: not at all, 2: a little, 3: quite, 4: a lot) are assigned according to the patient's responses to the item, only in items 29 and 30 are they evaluated with a score of 1 to 7 (1: dreadful, 7: excellent). The scores obtained are standardized to 0-100.

OTHER OUTCOMES:
TROP-2 positive rate | Baseline
  Determined centrally on most recent archival tumor samples collected at baseline. Percentage/proportion of patients considered positive for the expression of TROP-2 gene. Strong complete membranous staining in >5% of cells was considered positive.

CONTACTS AND LOCATIONS:
Overall Officials: Alejandro García-Alvarez, M.D.; Ph.D., Study Chair — Hospital Universitario Vall d´Hebron; Jaume Capdevila, M.D.; Ph.D., Study Chair — Hospital Universitario Vall d´Hebron
Locations (11):
- Spain (11):
  - Hospital Universitari Vall d'Hebron, Barcelona
  - Complexo Hospitalario Universitario de Ferrol, Ferrol
  - Institut Catala d´Oncologia (ICO) -Hospitalet, Hospitalet de Llobregat (Barcelona)
  - Hospital Clínico San Carlos, Madrid
  - Hospital Universitario la Paz, Madrid
  - Hospital Universitario Ramón y Cajal, Madrid
  - MD Anderson Cancer Center Madrid, Madrid
  - Hospital General Universitario Morales Meseguer, Murcia
  - Hospital Universitario Central de Asturias, Oviedo
  - H.U. Marqués de Valdecilla, Santander
  - Hospital Universitario Miguel Servet, Zaragoza

IPD SHARING:
Plan to Share IPD: Undecided
Provided upon reasonable request. All compiled or single patient data supporting the results will be publicly available.